CLINICAL TRIAL: NCT01227161
Title: New Formula for Selection of Proper Size of ETT in Children: Ultrasonographic Examination
Brief Title: New Formula for Selection of Proper Size of Endotracheal Tube (ETT) in Children: Ultrasonographic Examination
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Hae-Keum Kim / Professor, Department of Anesthesiology and Pain Medicine, Severance Hospital
Other Study IDs: 4-2009-0723
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Elective Urological Surgery
Keywords: ASA I-II children between the age 0-7; general anesthesia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasonography children: American Society of Anesthesiologists (ASA) I-II children between the age 0-7, undergoing elective urological surgery, such as inguinal hernia repair, orchiopexy, ureteroneocystostomy

SUMMARY:
Choosing the adequate size of endotracheal tube(ETT) in pediatric patients is important in all anesthesiologists, pediatricians, and critical care specialists. Inadequate ETT size will results in soft tissue injury to trachea by means of the pressure, insufficient ventilation, and aspiration, therefore choosing the adequate ETT size has very important clinical aspect.

DETAILED DESCRIPTION:
Choosing the adequate size of endotracheal tube(ETT) in pediatric patients is important in all anesthesiologists, pediatricians, and critical care specialists. Inadequate ETT size will results in soft tissue injury to trachea by means of the pressure, insufficient ventilation, and aspiration, therefore choosing the adequate ETT size has very important clinical aspect.

Subglottis is the narrowest portion of upper airway. Thus, ETT size should be determined according to the subglottic diameter. Several conventional methods are available to determine ETT size. These methods are based on the demographic data of patient, such as age, weight, height, but could not be customized for each patient. Ultrasonography (US) is one of the most accurate method to measure the subglottic diameter. Also, US is quick, easy to perform, and non-invasive measure. The investigators tried to measure the exact subglottic diameter with US and analyze the correlation of the diameter and demographical data. Furthermore, the investigators will try to develop the equation that could determine the adequate ETT size based on demographical data, instead of actually measuring the subglottic diameter using US.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing elective urological surgeries

Exclusion Criteria:

* children with anatomical airway problem or prematurely delivered children

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: University Hospital (Severance Hospital, Seoul, S.Korea)
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea